CLINICAL TRIAL: NCT01258959
Title: Anaesthesia for Ophthalmic Surgery: How "Retro" is the Peribulbar Block?
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Paul McHardy, Sunnybrook Health Science Centre
Other Study IDs: Retro-Parabulbar
Record Dates: First submitted 2010-12-08; First posted 2010-12-13 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2010-12

CONDITIONS: Ophthalmic Surgery; Parabulbar Block
Keywords: Ultrasound, retrobulbar, parabulbar, ophthalmic surgery.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ophthalmic surgery patients: Patients (men and women) of at least 18 years of age undergoing an ophthalmic procedure on the posterior section of the eye under local anaesthesia, i.e. with a peribulbar block. Inclusion and exclusion criteria for the study are the same as for the peribulbar anaesthesia.
  Interventions: Procedure: Ultrasound detection of local anesthetics spread

INTERVENTIONS:
Procedure: Ultrasound detection of local anesthetics spread — During the parabulbar injection the ultrasound operator experienced in ultrasound guided retrobulbar block will assess whether there is spread of local anaesthetic in the central cone just behind the sclera (yes or no). The anaesthesist performing the block will be blinded to the ultrasound visualized spread of local anaesthetic.

SUMMARY:
Ophthalmic surgery on the posterior section of the eye can either be performed under general anaesthesia or under local aneasthesia. The local anaesthesia is performed by injecting local anaesthetics behind the eye. There are two techniques: Either the needle is placed into the muscle cone formed by the four recti muscles - this is called intraconal or retrobulbar block, or the needle is placed outside of the muscle cone - this would be called extraconal or peribulbar. In our hospital the investigators usually perform the peribulbar block since it is easier to perform and has a smaller risk to injure the eye. The investigators however realize that the parabulbar block is sometimes very efficient and sometimes not, thus requiring a second or third injection. Now investigators are able to visualize where the local anaesthetics spreads with the help of ultrasound imaging. The aim of the study is to observe and to describe the incidence of intraconal spread of local anaesthetics when a peribulbar block is performed.

ELIGIBILITY:
Inclusion Criteria:

-informed consent

Exclusion Criteria:

* coagulation disorder
* INR over 1.5 and/or a platelet count less than 75 X 109/L,
* pathological myopia,
* inability of the patient to lie down for the operation for more than 2 hours
* lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 consecutive patients (men and women) of at least 18 years of age undergoing an ophthalmic procedure on the posterior section of the eye under local anaesthesia, i.e. with a peribulbar block.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Incidence of detectable retrobulbar spread of local anaesthetics during peribulbar injection. | At start (During peribulbar injection)
  The outcome measure is the description of the spread of local anesthetics during the injection of the drug via the parabulbar needle.

SECONDARY OUTCOMES:
Assessment of block quality | 20 Minutes after block
  Assessment of the block quality by ophthalmic surgeon just before surgery starts and at least 20 minutes after the block: complete akinesia and anaesthesia or partial akinesia/anaesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Science Centres, Toronto, Ontario, Canada

REFERENCES:
- [Background] Luyet C, Eichenberger U, Moriggl B, Remonda L, Greif R. Real-time visualization of ultrasound-guided retrobulbar blockade: an imaging study. Br J Anaesth. 2008 Dec;101(6):855-9. doi: 10.1093/bja/aen293. Epub 2008 Oct 23. PMID 18948389
- [Background] Ripart J, Lefrant JY, de La Coussaye JE, Prat-Pradal D, Vivien B, Eledjam JJ. Peribulbar versus retrobulbar anesthesia for ophthalmic surgery: an anatomical comparison of extraconal and intraconal injections. Anesthesiology. 2001 Jan;94(1):56-62. doi: 10.1097/00000542-200101000-00013. PMID 11135722
- [Background] Ropo A, Nikki P, Ruusuvaara P, Kivisaari L. Comparison of retrobulbar and periocular injections of lignocaine by computerised tomography. Br J Ophthalmol. 1991 Jul;75(7):417-20. doi: 10.1136/bjo.75.7.417. PMID 1854695